CLINICAL TRIAL: NCT06108050
Title: A Phase 1, First-in-human, Open-label, Multicenter Study of JZP898 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced or Metastatic Solid Tumors
Brief Title: JZP898 Intravenous Infusion as Monotherapy and Combination With Pembrolizumab in Adults With Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JZP898-101; KEYNOTE-F62 (Other: Merck Sharp & Dohme LLC); MK-3475-F62 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Advanced Solid Tumor; Metastatic Solid Tumor; JZP898
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A1 Dose Exploration: JZP898 monotherapy (Experimental)
  Interventions: Drug: JZP898
- Part A2 Dose Exploration: JZP898 in combination with pembrolizumab (Experimental)
  Interventions: Drug: JZP898; Drug: Pembrolizumab
- Part B Combination Expansion: JZP898 in combination with pembrolizumab (Experimental)
  Interventions: Drug: JZP898; Drug: Pembrolizumab

INTERVENTIONS:
Drug: JZP898 — Investigational drug monotherapy
Drug: Pembrolizumab — Anti-PD1 antibody
  Arms: Part A2 Dose Exploration: JZP898 in combination with pembrolizumab; Part B Combination Expansion: JZP898 in combination with pembrolizumab

SUMMARY:
This Phase 1 first-in-human study will investigate the safety, tolerability, pharmacokinetics (PK), immunogenicity, and preliminary antitumor activity of JZP898 monotherapy as well as JZP898 in combination with pembrolizumab in adult participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Two-part study: Part A Dose Exploration (Parts A1 and A2) and Part B Combination Expansion.

Part A Dose Exploration:

* Part A1 - a monotherapy dose exploration to determine the monotherapy recommended dose and/or maximum tolerated dose (MTD) (or highest cleared dose level) and safety profile of JZP898.
* Part A2 - a combination dose exploration of JZP898 plus pembrolizumab to determine the CombiRD (combination recommended dose for expansion).

Part B Combination Expansion:

* Part B - combination expansion using a basket design to evaluate clinical antitumor activity and safety profile of JZP898 in combination with pembrolizumab at the CombiRD identified in Part A2.

ELIGIBILITY:
Inclusion Criteria

* Adult ≥ 18 years of age
* Histological or cytological diagnosis of advanced or metastatic solid tumor.

  1. Previously treated participants with solid tumors that are amenable to CPI therapy (eg. NSCLC, melanoma, HNSCC, RCC, HCC, gastroesophageal carcinomas, UC, or CRC [MSI-H]) for whom, in the opinion of the investigator, there is no SoC available to convey clinical benefit.
  2. Parts A2 and B: previously-treated (≥ 1 line of prior anticancer therapy) participants with select tumor types (NSCLC, HNSCC, melanomas, RCC, and UC) who have progressed on/after prior CPI therapy based on investigator assessment per RECIST version 1.1.
* Participants in select tumor types:

  1. NSCLC: eligible for platinum-based therapy and received platinum-based therapy prior to inclusion in the study.
  2. HNSCC: eligible for platinum therapy and received platinum-based therapy prior to inclusion in this study.
  3. Melanoma with known BRAFv600 mutation: received BRAF/MEKi therapy before this study.
* ECOG score of 0 to 1.
* Measurable disease per RECIST version 1.1 criteria.
* Parts A1 and A2 only: willing to consent to mandatory tumor biopsies (both pretreatment and post-treatment with JZP898) unless medically infeasible
* Adequate organ and bone marrow function as indicated by the following laboratory values (within 4 weeks prior to starting the study interventions)
* Men and women of reproductive potential to observe highly effective birth control for the duration of treatment and for 4 months following the last dose of study drug;
* Additional criteria may apply

Exclusion Criteria

* Unresolved toxicities from previous therapy that is > Grade 1.
* Hypersensitivity to mAb, IFNα, or study intervention components.
* Primary CNS tumor or symptomatic CNS metastases.
* Have a second primary malignancy treated within the previous 2 years (exceptions: non-metastatic, non-melanomatous skin cancers, carcinoma in-situ, and melanoma in-situ).
* Active autoimmune disease (in the last 2 years) requiring systemic steroids or immunosuppressive agents.
* Active or history of pneumonitis (noninfectious) or interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Any history of suicidal behavior or any suicidal ideation
* Clinically significant ischemic/hemorrhagic cerebrovascular accident/stroke and/or clinically significant active cardiovascular disease
* Received any anticancer therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug
* Received prior radiotherapy within 2 weeks of the first dose of study drug or have had a history of radiation pneumonitis
* Major surgery within 2 weeks prior to the first dose of study intervention.
* Participant is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Had a stem cell/solid organ transplant.
* Receipt of prior IFNα therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities in Monotherapy and Combination Therapy | Up to 36 months
Incidence of TEAEs and SAEs in Monotherapy and Combination Therapy | Up to 36 months
Incidence of dose interruptions, discontinuation, and reductions due to TEAEs in Monotherapy and Combination Therapy | Up to 36 months
Objective Response Rate (ORR) As Assessed by the Investigator In Combination Therapy | Up to 36 months

SECONDARY OUTCOMES:
Pharmacokinetic Parameter: Maximum Concentration (Cmax) of JZP898 in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Time to Maximum Concentration (Tmax) of JZP898 in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Terminal Elimination Half-life (t½) of JZP898 in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Area Under the Concentration-Time Curve (AUC) of JZP898 in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Clearance (CL) of JZP898 in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Volume of Distribution (V) of JZP898 in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Activated IFNα-to-JZP898 Ratio in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Accumulation ratio for Cmax in Monotherapy and Combination Therapy | Up to 36 months
Pharmacokinetic Parameter: Accumulation Ratio for AUC in Monotherapy and Combination Therapy | Up to 36 months
ORR As Assessed by the Investigator in Monotherapy | Up to 36 months
Duration of Response (DoR) As Assessed by the Investigator | Up to 36 months
Disease Control Rate (DCR) As Assessed by the Investigator | Up to 36 months
Progression-free Survival (PFS) As Assessed by the Investigator | Up to 36 months
Overall Survival (OS) | Up to 36 months
Incidence of ADAs towards JZP898 | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Orlando, Florida
  - Duke University Medical Center - Duke Cancer Institute, Durham, North Carolina
  - Sidney Kimmel Cancer Center at Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No